CLINICAL TRIAL: NCT01192048
Title: Genetic Testing of Individuals and Families With Congenital Heart Disease
Brief Title: Genetics of Congenital Heart Disease
Status: Recruiting | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Vidu Garg, Director and Professor, Nationwide Children's Hospital
Other Study IDs: IRB09-00339; R01HL109758 (NIH)
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; birth defect; genetics; gene; DNA; direct sequencing; microarray; single nucleotide polymorphism; whole genome array comparative genomic hybridization; chromosomal copy number change; nucleotide sequence variation; exome sequencing; whole exome sequencing; whole genome sequencing
MeSH Terms: conditions — Heart Defects, Congenital; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected in vacuum tubes containing acid citrate dextrose (ACD). Lymphocytes from blood drawn in appropriate anticoagulant (ACD) may be stored for subsequent immortalization. DNA will be extracted from these samples for analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Subjects: Individuals with Congenital Heart Disease and family members with or without Congenital Heart Disease. A blood sample collection will be required for all study participants.
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Blood sample collection for direct sequencing, microarray, single nucleotide polymorphism, whole-genome array comparative genomic hybridization DNA analyses, and/or whole exome or genome sequencing.

SUMMARY:
Congenital heart disease (CHD) is the most common type of birth defect but the cause for the majority of cardiac birth defects remains unknown. Numerous epidemiologic studies have demonstrated evidence that genetic factors likely play a contributory, if not causative, role in CHD. While numerous genes have been identified by us and other investigators using traditional genetic approaches, these genes account for a minority of the non-syndromic CHDs. Therefore, we are now utilizing whole genome sequencing (WGS), with the addition of more traditional genetic techniques such as chromosomal microarray or traditional linkage analysis, to identify genetic causes of familial and isolated CHD. With WGS we are able to sequence all of the genetic material of an individual and apply different data analysis techniques based on whether we are analyzing a multiplex family or a cohort of trios (mother, father and child with CHD) with a specific isolated CHD. Therefore, WGS is a robust method for identification of novel genetic causes of CHD which will have important diagnostic and therapeutic consequences for these children.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is the most common type of birth defect, but the etiology of CHD remains largely unknown. Genetic causes have been discovered for both syndromic and non-syndromic CHD utilizing several genetic approaches (Yasuhara and Garg, 2021). The majority of these genetic causes have found by studying large families with autosomal dominant congenital heart disease and my laboratory has successfully used this methodology in the past (Garg, 2003; Garg 2005; Pan, 2009; Bennett, 2022). Although these positional cloning approaches are very powerful, they are limited by rare nature of multi-generation pedigrees and are limited to milder forms of CHD that have allowed for the generation of large kindreds.

The other method that has traditionally been utilized to identify genetic causes of CHD is the screening of large populations of children with sporadic (non-familial) cases of CHD for genetic abnormalities (nucleotide sequence variations in candidate genes for CHD or for chromosomal copy number changes that involve CHD-candidate genes). This work has been tedious as a large number of candidate genes have been implicated as potentially responsible for CHD in humans (Choudhury and Garg, 2022). Although this approach has been successful (Schluterman, 2007; Maitra, 2010; Chang, 2013; Bonachea, 2014), it is also limited to the candidate gene lists.

Whole exome sequencing (WES) is a next-generation sequencing technology that allows for the sequencing of all of the expressed genes. Our group, in addition to several others (LaHaye, 2016; Gordon, 2022), has been utilizing WES technology for CHD gene discovery. Our group has progressed to utilizing whole genome sequencing (WGS), a next-generation sequencing technology that allows for the sequencing of all genetic material (including genomic regions that are not sequenced in WES), in our analysis for CHD gene discovery. Therefore, these sequencing methods can be applied to multiplex families and cohorts of sporadic cases to identify genetic causes of CHD in an unbiased manner. Genomic sequencing is dependent on the technical and bioinformatics prowess of the personnel running the sequencing and the controlling the data pipeline. The Institute of Genomic Medicine at Nationwide Children's Hospital (NCH) is both technically skilled and have developed their own powerful data pipeline (Kelly, 2015). WGS is a powerful genetic tool that can be used in isolation or in conjunction with other types of genetic analysis to increase the yield of these investigations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of Congenital Heart Disease or be related to individuals with Congenital Heart Disease.

Exclusion Criteria:

* Healthy individuals unrelated to those with Congenital Heart Disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: cardiology clinic sample, community sample
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-12; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of novel genetic contributors to congenital heart defects | up to 3 years, from date of genetic analysis to completion of genetic data analysis or identification of novel genetic contributors, whichever comes first
  Novel genetic abnormalities that are found to be associated with congenital heart defects in humans

CONTACTS AND LOCATIONS:
Overall Officials: Vidu Garg, MD, Principal Investigator — The Research Institute at Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Pan H, Richards AA, Zhu X, Joglar JA, Yin HL, Garg V. A novel mutation in LAMIN A/C is associated with isolated early-onset atrial fibrillation and progressive atrioventricular block followed by cardiomyopathy and sudden cardiac death. Heart Rhythm. 2009 May;6(5):707-10. doi: 10.1016/j.hrthm.2009.01.037. Epub 2009 Feb 4. No abstract available. PMID 19328042
- [Background] Maitra M, Koenig SN, Srivastava D, Garg V. Identification of GATA6 sequence variants in patients with congenital heart defects. Pediatr Res. 2010 Oct;68(4):281-5. doi: 10.1203/PDR.0b013e3181ed17e4. PMID 20581743
- [Background] Schluterman MK, Krysiak AE, Kathiriya IS, Abate N, Chandalia M, Srivastava D, Garg V. Screening and biochemical analysis of GATA4 sequence variations identified in patients with congenital heart disease. Am J Med Genet A. 2007 Apr 15;143A(8):817-23. doi: 10.1002/ajmg.a.31652. PMID 17352393
- [Background] Garg V, Muth AN, Ransom JF, Schluterman MK, Barnes R, King IN, Grossfeld PD, Srivastava D. Mutations in NOTCH1 cause aortic valve disease. Nature. 2005 Sep 8;437(7056):270-4. doi: 10.1038/nature03940. Epub 2005 Jul 17. PMID 16025100
- [Background] Garg V, Kathiriya IS, Barnes R, Schluterman MK, King IN, Butler CA, Rothrock CR, Eapen RS, Hirayama-Yamada K, Joo K, Matsuoka R, Cohen JC, Srivastava D. GATA4 mutations cause human congenital heart defects and reveal an interaction with TBX5. Nature. 2003 Jul 24;424(6947):443-7. doi: 10.1038/nature01827. Epub 2003 Jul 6. PMID 12845333
- [Background] Bonachea EM, Chang SW, Zender G, LaHaye S, Fitzgerald-Butt S, McBride KL, Garg V. Rare GATA5 sequence variants identified in individuals with bicuspid aortic valve. Pediatr Res. 2014 Aug;76(2):211-6. doi: 10.1038/pr.2014.67. Epub 2014 May 5. PMID 24796370
- [Background] Bonachea EM, Zender G, White P, Corsmeier D, Newsom D, Fitzgerald-Butt S, Garg V, McBride KL. Use of a targeted, combinatorial next-generation sequencing approach for the study of bicuspid aortic valve. BMC Med Genomics. 2014 Sep 26;7:56. doi: 10.1186/1755-8794-7-56. PMID 25260786
- [Background] LaHaye S, Corsmeier D, Basu M, Bowman JL, Fitzgerald-Butt S, Zender G, Bosse K, McBride KL, White P, Garg V. Utilization of Whole Exome Sequencing to Identify Causative Mutations in Familial Congenital Heart Disease. Circ Cardiovasc Genet. 2016 Aug;9(4):320-9. doi: 10.1161/CIRCGENETICS.115.001324. Epub 2016 Jul 14. PMID 27418595
- [Background] Bennett JS, Gordon DM, Majumdar U, Lawrence PJ, Matos-Nieves A, Myers K, Kamp AN, Leonard JC, McBride KL, White P, Garg V. Use of machine learning to classify high-risk variants of uncertain significance in lamin A/C cardiac disease. Heart Rhythm. 2022 Apr;19(4):676-685. doi: 10.1016/j.hrthm.2021.12.019. Epub 2021 Dec 24. PMID 34958940
- [Background] Yasuhara J, Garg V. Genetics of congenital heart disease: a narrative review of recent advances and clinical implications. Transl Pediatr. 2021 Sep;10(9):2366-2386. doi: 10.21037/tp-21-297. PMID 34733677
- [Background] Choudhury TZ, Garg V. Molecular genetic mechanisms of congenital heart disease. Curr Opin Genet Dev. 2022 Aug;75:101949. doi: 10.1016/j.gde.2022.101949. Epub 2022 Jul 8. PMID 35816939
- [Background] Chang SW, Mislankar M, Misra C, Huang N, Dajusta DG, Harrison SM, McBride KL, Baker LA, Garg V. Genetic abnormalities in FOXP1 are associated with congenital heart defects. Hum Mutat. 2013 Sep;34(9):1226-30. doi: 10.1002/humu.22366. Epub 2013 Jul 11. PMID 23766104
- [Background] Yasuhara J, Manivannan SN, Majumdar U, Gordon DM, Lawrence PJ, Aljuhani M, Myers K, Stiver C, Bigelow AM, Galantowicz M, Yamagishi H, McBride KL, White P, Garg V. Novel pathogenic GATA6 variant associated with congenital heart disease, diabetes mellitus and necrotizing enterocolitis. Pediatr Res. 2024 Jan;95(1):146-155. doi: 10.1038/s41390-023-02811-y. Epub 2023 Sep 12. PMID 37700164
- [Background] Gordon DM, Cunningham D, Zender G, Lawrence PJ, Penaloza JS, Lin H, Fitzgerald-Butt SM, Myers K, Duong T, Corsmeier DJ, Gaither JB, Kuck HC, Wijeratne S, Moreland B, Kelly BJ; Baylor-Johns Hopkins Center for Mendelian Genomics; Garg V, White P, McBride KL. Exome sequencing in multiplex families with left-sided cardiac defects has high yield for disease gene discovery. PLoS Genet. 2022 Jun 23;18(6):e1010236. doi: 10.1371/journal.pgen.1010236. eCollection 2022 Jun. PMID 35737725
- [Background] Manivannan SN, Darouich S, Masmoudi A, Gordon D, Zender G, Han Z, Fitzgerald-Butt S, White P, McBride KL, Kharrat M, Garg V. Novel frameshift variant in MYL2 reveals molecular differences between dominant and recessive forms of hypertrophic cardiomyopathy. PLoS Genet. 2020 May 26;16(5):e1008639. doi: 10.1371/journal.pgen.1008639. eCollection 2020 May. PMID 32453731